CLINICAL TRIAL: NCT06584006
Title: A Phase II, Single-Center, Randomized Controlled Clinical Trial Evaluating the Efficacy of Thymalfasin and Recombinant Human Interleukin-2 Injections in Treating Lymphocytopenia in Patients With Malignant Hematological Tumors
Brief Title: Thymalfasin and Recombinant Human IL-2 Injections in Treating Lymphocytopenia for Patients With Malignant Hematological Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Zhijuan Lin, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-12
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hematological Malignancy; Lymphocytopenia
MeSH Terms: conditions — Hematologic Neoplasms; Lymphopenia | interventions — Thymalfasin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combination Therapy Group (Experimental): Thymalfasin for injection in combination with Recombinant Human Interleukin-2 Injections
  Interventions: Drug: Thymalfasin for injection in combination with Recombinant Human Interleukin-2 Injections
- Monotherapy Group (Experimental): Recombinant Human Interleukin-2 Injections as a monotherapy
  Interventions: Drug: Recombinant Human Interleukin-2 Injections
- Control Group (No Intervention): non-intervention

INTERVENTIONS:
Drug: Thymalfasin for injection in combination with Recombinant Human Interleukin-2 Injections — Thymalfasin for injection 1.6mg subcutaneous injection once daily (qd) for 7 days, and Recombinant Human Interleukin-2 Injections 1 million units subcutaneous injection qd for 7 days.
  Other Names: Combination Therapy Group
  Arms: Combination Therapy Group
Drug: Recombinant Human Interleukin-2 Injections — Recombinant Human Interleukin-2 Injections 1 million units subcutaneous injection qd for 7 days.
  Other Names: Monotherapy Group
  Arms: Monotherapy Group

SUMMARY:
To evaluate the efficacy and safety of Thymalfasin for injection in combination with Recombinant Human Interleukin-2 Injections in the treatment of lymphocytopenia in patients with malignant hematological tumors

DETAILED DESCRIPTION:
A prospective, randomized controlled study is proposed to evaluate the efficacy and safety of Thymalfasin for injection in combination with Recombinant Human Interleukin-2 Injections, Recombinant Human Interleukin-2 Injections as a monotherapy, and a non-intervention group. Follow-up observations will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed myeloid, B lymphocyte, and plasma cell-derived malignant hematological tumors.
2. Lymphocyte count ≤ 0.8×109/L or CD4+T cell count ≤ 0.35×109/L.
3. Age ≥ 18 years, both male and female, with an expected survival period of more than 3 months.
4. Estimated creatinine clearance rate ≥ 30 mL/min.
5. AST and ALT ≤ 3.0 x ULN. Bilirubin ≤ 1.5 x ULN.
6. ECOG ≤ 2.
7. Able to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. Active autoimmune disease.
2. Patients considered to have a malignant T-cell clone.
3. Within 8 days after chemotherapy for lymphoma and within 14 days after chemotherapy for AML.
4. Tumor involvement in the bone marrow leading to hematopoietic suppression (neutrophils <1.0×10^9/L, HB<70g/L, PLT<50×10^9/L).
5. HIV-positive patients and/or active HBV or HCV infection (as evidenced by positive HBV-DNA and HCV-RNA test records).
6. Patients with chronic respiratory diseases requiring continuous oxygen, or with significant past medical history of kidney, neurological, psychiatric, endocrine, metabolic, immune, hepatic, cardiovascular diseases.
7. Immunosuppressive treatment (such as cyclosporine, corticosteroids, ruxolitinib, JAK1/2 inhibitors, etc.) within the past 5 days.
8. Psychiatric disorders that would interfere with study participation.
9. Patients who have undergone allogeneic hematopoietic stem cell transplantation.
10. Consideration of allergy to Thymalfasin or Interleukin-2.
11. Any other condition that the researcher believes makes the patient unsuitable for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Lymphocyte count and its subgroup count | Up to 36 months
  Dynamic changes in lymphocyte count and its subgroup count

SECONDARY OUTCOMES:
NK cells | Up to 36 months
  Changes in NK cells
Infection | Up to 36 months
  Incidence of infections
Treatment interruption | Up to 36 months
  Rate of treatment interruption or delay.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijuan Lin, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Zhijuan Lin, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No